A randomized trial evaluating single fraction stereotactic versus standard multi-fraction radiotherapy for patients diagnosed with bone metastases for effective palliation of symptoms.

# 1. OBJECTIVES:

- a. Primary objective (phase II): evaluate single fraction stereotactic regimen for pain response in terms of time to failure, defined as the first occurrence of any of the following events:
  - i. worsening in pain score by at least 2 categories by MDASI survey,
- b. Primary objective (phase III): to evaluate the pain response at 3 months in terms of pain response by a decrease in 2 categories by MDASI survey and narcotics use as defined by international pain consensus criteria.
- c. Secondary objective: report outcomes
  - i. Compare narcotics/opioid use compared to baseline, ≥ 50% increase in dose of opioid/narcotic medication,
  - ii. re-irradiation,
  - iii. radiographic disease progression or development of pathologic fracture from disease progression
  - iv. Prospectively report pain, quality of life, and symptoms using MDASI assessment tool to measure pain response
  - v. Report acute (skin, fatigue, flare reaction) and long term (sclerosis, bone ossification, bone fracture rate) toxicity associated with treatment.
  - vi. Report local control and overall survival
  - vii. Report rate of salvage surgery

### 2. BACKGROUND:

a. Radiation therapy is commonly utilized to effectively palliate symptomatic bone metastases, 50%-80% of patients experience improvement in the pain and 20%-50% report complete pain relief (1, 2). However, the optimal fractionation scheme to produce durable pain relief is still being studied. Historically, clinical trials have compared efficacy of varying dose-fractionation in alleviating symptoms. Ratanatharathorn et al. concluded in their analysis that higher dose fractionated treatments produced better pain outcomes compared to lower-dose regimens (3, Ratanatharathorn). Contrary to this, McQuay et al. in their summary determined no difference in efficacy between different fractionation or dose response in the total dose delivered for painful bone metastases (4, McQuay). In the meta-analysis performed by Wu et al (5, Wu) the authors compared pain relief among various dose-fractionation schedules of localized radiotherapy (RT) in the treatment of painful bone metastases. They concluded among the randomized trials, there was no significant difference in overall pain

relief or dose response relationship between single and multi-fraction palliative RT for bone metastases.

In the last two decades, multiple randomized trials have compared the efficacy of various dose-fractionation in achieving durable pain relief in patients diagnosed with bone metastases. A randomized trial, RTOG 9714 investigated whether 8 Gy delivered in a single fraction provided pain and narcotic relief equivalent to the standard 30 Gy in 10 fractions. The study demonstrated both regimens were equivalent in terms of pain and narcotic relief, and well tolerated with few adverse effects. The shorter 8 Gy arm had a higher re-treatment rate but with less acute toxicity than the longer 30 Gy arm (6, Hartsell). However, the Trans-Tasman Radiation Oncology Group (TROG 96.05) was a randomized trial which demonstrated 8 Gy in a single fraction was not as effective as 20 Gy in 5 fractions; the overall response rate and time to treatment failure were inferior (7, Roos). The re-treatment rate has been reported to be higher in patients treated by single fraction radiotherapy; this could be due to the decrease in durability of pain response related to the lower dose equivalent (8, Sze).

A single delivery of higher dose of radiation treatment can be advantageous in regards to patient convenience and cost effectiveness as long as it can provide durable pain control. The optimal single fraction dose required to achieve pain control is still unknown and not determined from current clinical trials. Gaze et al demonstrated and overall pain response rate of 84% and complete pain response rate of 34% with delivery of a single fraction of 10 Gy (9, Gaze) for patients with osseous metastases. Higher doses of 12 Gy and 15 Gy have demonstrated a dose response of increased overall pain response of 86% and complete pain response in 57% of patients (10, Kagei). Radiosurgery doses of >16 Gy has been shown to increase the probability of pain relief for patients with spine metastases by multiple institutions such as Henry Ford and University of Pittsburgh (11, 12, Ryu, Gerzten). Researchers at M.D. Anderson have demonstrated the use of single fraction SBRT with doses of 16-24 Gy for spinal metastases was safe and allowed patients to achieve durable local control (88% at 18 months) with few toxicities (13, Garg).

Multiple prospective randomized trials have investigated the efficacy of shorter versus longer fractionated radiation therapy courses for the treatment of painful bone metastases with conflicting results. Few studies prospectively address the relief of neuropathic pain, re-irradiation rates, fracture rates and prospective quality of life endpoints. In this study, we propose to deliver a dose escalated single fraction (12 Gy or 16 Gy) regimen compared to the standard 20 Gy in 5 fractions to report the safest optimal hypofractionated regimen in providing durable symptomatic relief.

# 3. SCIENTIFIC RATIONALE:

a. This study aims to prospectively evaluate the optimal radiation therapy dose to provide durable pain relief, assess patients' quality of life, narcotics use after radiation therapy, outcome, and toxicity. The goal of this prospective randomized trial is to radiate patients with mechanically stable, painful bone metastases effectively to provide quick palliation of pain. The hypothesis is rapid delivery of dose escalated hypofractionated radiotherapy for bone metastases effectively improves pain and results in durable pain control.

#### 4. PATIENT ELIGIBILITY

### a. INCLUSION:

- i. Patients with a pathologic diagnosis of malignancy
- ii. Patients with any radiographic evidence of bone metastases, including plain x-ray, bone scan, CT scan, MRI, or PET scan
- iii. Patients with pain or dysathesia
- iv. Patients with a life expectancy of more than 3 months
- v. Patients able to complete pain assessment and quality of life surveys
- vi. Patients with multiple osseous sites are eligible; however should not treat more than 3 separate radiation treatment fields concurrently.
- vii. Patients with surgery for osseous metastases allowed.

#### b. EXCLUSION:

- i. Patients with prior radiation therapy to the treatment site
- ii. Patients with a current, untreated spinal cord compression
- iii. Patients with a radiographic or pathologic fracture to the treatment site
- iv. Patients with painful metastases to hands and feet that need to be radiated on protocol
- v. Patients previously treated with radioactive isotope (e.g. Sr89) within 30 days of randomization

### 5. PRE-TREATMENT EVALUATION:

- a. The workup will include physical examination, radiographic evidence of metastases with either x-ray, bone scan, CT scan or MRI, and pathologic confirmation of malignancy per MDACC standard of care.
- b. All eligible patients will be enrolled after completion of the eligibility checklist.
- c. Use of pain medications (narcotic/opioids/NSAIDs) will be evaluated.

# 6. TREATMENT PLAN:

- a. Patients will be randomized to receive radiation therapy to:
  - i. Arm 1: the standard hypofractionated regimen of 3 Gy x 10 fractions
  - ii. Arm 2: 12 Gy x 1 fraction or 16 Gy x 1 fractions adaptively depending on the size of the metastases or gross tumor volume (GTV).
- b. Patients will undergo CT simulation and either 2-D or 3-D treatment planning for radiation therapy.

- c. Patients can be treated with 2-D, 3-D, or intensity modulated radiation therapy (IMRT)
- d. Patients will be treated with on board imaging (OBI) using KV, MV x-rays, cone beam CT or CT on rails per standard of care.
- e. Patients will be treated with 4-20 MV photon beam, 5-20 MeV electron beam, or 200 MeV-300 MeV proton beam.
- f. More than 1 osseous site may be included into one radiation treatment field.

# 7. EVALUATION DURING STUDY:

- a. All patients will be evaluated by the radiation oncologist during radiation treatment
- b. If surgical intervention is necessary, the patients will be evaluated by the treating surgeon
- c. After start of treatment, all patients will be followed by phone calls within 7-14 days, and at + 1 month (+/- 1 week) and then with clinic visits at months 3, 6, 9, 12 (+/- 4 weeks for each visit) and every 3 to 6 month intervals thereafter (until death) by either the radiation oncology or orthopedic team to evaluate toxicity. The validated surveys (MDASI) will be completed at baseline prior to radiation and at each follow up interval/appointments. The patient medical record number will be placed on the survey before it is given to the patient for completion. The surveys may be filled out in person or by mail.
- d. Patients will report their symptom measures with validated quality of life instrument MDASI index. The M.D. Anderson Symptom Inventory (MDASI) is a multi-symptom patient reported outcome measure evaluating 13 core symptom items interfering with patients' daily life (Appendix B).
- e. We will also prospectively report the narcotics/NSAIDs utilization and outcome at each follow-up interval after radiation therapy.

### 8. EVALUATION OF TOXICITY:

- a. During radiotherapy, the patient will be examined weekly and acute reactions recorded.
- b. Toxicity occurring after 3 months of radiation therapy; these will be evaluated and documented using NCI CTCAE version 4.03 (Appendix A).

#### 9. CRITERIA FOR RESPONSE:

- a. The response to treatment will be determined by both radiographic scans and symptoms reported.
- b. Complete pain relief is defined as average pain score of 0 for two consecutive analysis periods.
- c. The time to maximal relief of pain is defined from the first day of irradiation until the lowest pain score after radiation therapy.

- d. Treatment failure is defined as worsening of pain by at least two categories, >50% increase in dose of opioid/narcotic medications, re-irradiation for pain or disease progression, progression or development of pathologic fracture from disease progression.
- e. Any patient with progressive pain in the radiated area will have work up which include radiographic scans to evaluate for bone stability and pathologic fracture per standard of care.

#### 10. <u>RE-TREATMENT:</u>

- a. Response and pain relief from radiation therapy may take several weeks; therefore patients should not be re-irradiated for at least 4 weeks after completion of radiation. Dose and fractionation are left to the discretion of the treating radiation oncologist.
- b. Surgical intervention for treatment failures, bone instability, or fractures will be reported.

#### 11. STATISTICAL CONSIDERATIONS:

This is a phase II/III non-inferiority trial following the design suggestions of Korn et al. (14, Korn). The primary outcome for phase II part is treatment failure at 1 month, where treatment failure is as defined in section 1.0. We assume that time to treatment failure follows an exponential distribution for each treatment arm (standard radiation, hypofractionated radiation). We also assume that the standard radiation arm will have 25% of patients with treatment failure at 3 months, based on the study by the Bone Pain Trial Working Party (15, BPTWP). A hazard ratio of 1.5 implies that the hypofractionated radiation arm will have 35% of patients with treatment failure at 3 months. The primary outcome for phase III part is pain response rate at 3 months post randomization. We expect to enroll 10 patients per month.

#### Randomization

Patients will be randomized to standard or single fraction stereotactic radiation therapy using CORe. Randomization will be stratified by tumor size ( $\leq 4$  cm vs. > 4 cm), site of bony mets (extremities, pelvis, abdomen, head/neck, chest), and 1 vs > 1 site irradiated. We expect approximately 40% of patients will have bony mets in the extremities and approximately 35% will have bony mets in the pelvis. We expect the distribution of patients enrolling will approximately be 40% lung malignancy, 25% genitourinary malignancy, 15% breast malignancy, 10% multiple myeloma and 10% other malignancy. We will have a total of 14 stratification levels.

#### Phase II

We will test the following hypothesis:

 $H_0$ :  $\rho = 1.5$  vs.  $H_1$ :  $\rho = 1.0$ ,

where  $\rho$  is the hazard ratio (hypofractionated/standard) for time to treatment failure, as defined in section 1.0. A sample size of 150 patients (75 randomized to each treatment arm) will yield 90% power with a 1-sided significance level of 0.20 to reject the null hypothesis (H<sub>0</sub>) and conclude that hypofractionated treatment is not inferior to standard treatment in terms of time to treatment failure. We use a 1-sided significance level of 0.20 as recommended by Rubinstein et al. (16, Rubinstein) for phase II screening trials. This sample size will yield 110 events (i.e., treatment failures). It will take 15 months to enroll all the patients, and the maximum study duration is expected to be 22 months to observe the 110 events. The final analysis for phase II will be performed once we've observed 110 events, and we will suspend accrual while we wait for these events to occur. We will continue to phase III only if we reject H<sub>0</sub> at the 0.20 significance level.

#### Phase III

The patients enrolled in the phase III part of the study will be included in the phase III part of the study. In the Phase II trial, we have already enrolled and randomized 160 patients, therefore we are requesting to enroll another additional 50 patients to reach a total of 210 patients. We will enroll another 50 patients in total of 210 patients (105 randomized to each treatment arm), after the rejection of the  $H_0$  in the phase II part of the trial. The primary objective is to evaluate the pain response at 3 months by international pain consensus criteria after the additional 50 patients have been accrued, we will follow all patients for at least 3 months to assess the pain response. Assuming a 20% of the 3-month pain response rate for patients on MFRT arm, the 210 patients will ensure an 80% power to detect a 16% improvement in response rate (36%) with SBRT using a 1-sided 5% level test.

Pain response at 3 months is defined as reduction in pain score reported by MDASI at 2 points below baseline also taking into account narcotics use, as defined by International Pain Response Criteria.

This sample size calculation was performed using East 6 (Copyright © 2010, Cytel Inc., Cambridge, MA).

Toxicity Monitoring (phase II and phase III)

We will monitor the rate of radiation induced toxicity (skin dermatitis grade  $\geq 4$ , gastrointestinal (GI) grade  $\geq 3$ , genitourinary (GU) grade  $\geq 3$ ) by 12 months after the start of radiation therapy for the hypofractionated radiation therapy arm. We will enroll at least 25 patients and at most 105 patients on this treatment arm, and we will use the methods of Thall et al. (17, Thall et al.) to monitor the radiation induced toxicity rate.

We will stop enrolling patients on the hypofractionated radiation therapy arm if we have reason to believe that the rate of radiation induced toxicity for this arm is more than 10%.

We will actually monitor the time to radiation induced toxicity, because these toxicities may occur at any time from the start of radiation therapy. We will use the Clinical Trial Conduct website (<a href="https://biostatistics.mdanderson.org/ClinicalTrialConduct">https://biostatistics.mdanderson.org/ClinicalTrialConduct</a>) to monitor the toxicity stopping rule. This website is built and maintained by the Department of Biostatistics. The research staff will be trained by the study statistician in the use of the website to monitor the stopping rules, with an emphasis on the importance of updating toxicity outcomes and follow-up dates.

To obtain the operating characteristics for the stopping rule we simulated the trial 1000 times for various scenarios described in the table below. We assumed that patients are enrolled at the rate of 5 per month on the hypofractionated radiation therapy arm, that we would follow patients for 12 months, and that we will evaluate the stopping rule continually. The table below summarizes the operating characteristics of this stopping rule.

| Operating Characteristics for the Toxicity Monitoring Rule | | | | | | |
|---|---|---|---|---|---|---|
| Median time to | | | Sample Size | | | Avg Trial |
| radiation | 12-Month | Pr(Stop | | - | | Duration |
| induced toxicity | Toxicity Rate | Early) | P <sub>25</sub> | 25 Mean | P <sub>75</sub> | (Months) |
| (months) | | | | | | (IVIOTILIS) |
| 120 | 0.07 | < 0.001 | 105 | 105 | 105 | 33.2 |
| 60 | 0.13 | 0.113 | 105 | 103 | 105 | 32.8 |
| 40 | 0.19 | 0.667 | 77 | 89 | 105 | 30.1 |
| 30 | 0.24 | 0.949 | 60 | 73 | 85 | 26.9 |

At any point in the trial time to radiation induced toxicity can be calculated for each patient, with the time interval regarded as censored at the date of last follow-up if toxicity has not been observed for a patient. We will apply a Bayesian method for updating prior information with time to toxicity data observed to that time. We assume that the time to toxicity for each patient is exponentially distributed with a median of  $\lambda_S$  months for the standard treatment and a median of  $\lambda_S$  for the experimental treatment. Given the historical data we assume  $\lambda_S$  follows an inverse gamma distribution with mean 78.95 months and a standard deviation of 0.15 months. The middle 95% of this distribution is between 78.66 and 79.24 months. These parameters correspond to a 12-month toxicity rate between 9.064% and 10.035%. We assume  $\lambda_S$  follows an inverse gamma distribution with a mean of 78.95 months and a standard deviation of 15.0 months. The middle 95% of this distribution is between 54.87 and 113.32 months. These parameters correspond to a 12-month toxicity rate between 7.077% and 14.066%.

Since the goal of the study is to achieve a toxicity rate of less than 10% at 12 months, the trial will be stopped early if, based on the available data, Pr( $\lambda_E < \lambda_S$  | data from the trial) >0.90. This rule was chosen to achieve an approximately 0.10 early stopping probability if the true toxicity rate is 10%.

## Final Analysis

We will use descriptive statistics to summarize the demographic and clinical characteristics of patients by treatment arm.

We will use the methods of Gooley et al. (18, Gooley) to estimate the cumulative incidence of treatment failure for each treatment arm with death as a competing event, and we will estimate the percent of patients without treatment failure at 3, 6, and 12 months for each treatment arm with a 90% confidence interval.

We will use the methods of Fine and Gray (19, Fine and Gray) to model time to treatment failure with death as a competing event and test the hypotheses stated above for phase II and for phase III. We will also estimate the hazard ratio for treatment with a 90% confidence interval.

For the 3 month pain response rate, the Cochran-Mantel-Haenszel test stratified by stratification factors at randomization will used to test the difference between 2 treatment arms. Chi-squared test without adjusting for the stratification factors will also be performed as a secondary analysis.

We will use descriptive statistics and boxplots to summarize the score from the MDASI instrument at each assessment time. We will similarly summarize changes in scores for these instruments over time. We will use mixed effects regression methods with repeated measures and patient as a random effect to model instrument scores over time to test for treatment differences.

We will use the product limit estimator of Kaplan and Meier (20, Kaplan and Meier) to estimate overall survival and disease-free survival stratified by treatment arm. We will use Cox proportional hazards regression to model OS and DFS as a function of treatment arm, and we will estimate the hazard ratio for treatment with a 90 % confidence interval (21, Cox).

We will use descriptive statistics to summarize narcotics use and acute and long-term adverse events for each treatment arm.

We will use Fisher's exact test to compare treatment arms with respect to the rates of re-irradiation and salvage surgery.

# 12. Database:

Study data will be collected and managed using REDCap (Research Electronic Data Capture) electronic data capture tools hosted at MD Anderson. [ref 22] REDCap (<a href="www.project-redcap.org">www.project-redcap.org</a>) is a secure, web-based application with controlled access designed to support data capture for research studies, providing: 1) an intuitive interface for validated data entry; 2) audit trails for tracking data manipulation and export procedures; 3) automated export procedures for seamless downloads to common statistical packages; and 4) procedures for importing data from external sources. REDCap (<a href="https://redcap.mdanderson.org">https://redcap.mdanderson.org</a>) is hosted on a secure server by MD Anderson Cancer Center's Department of Research Information Systems & Technology Services. REDCap has undergone a Governance Risk & Compliance Assessment (05/14/14) by MD Anderson's Information Security Office and found to be compliant with HIPAA, Texas Administrative Codes 202-203, University of Texas Policy 165, federal regulations outlined in 21CFR Part 11, and UTMDACC Institutional Policy #ADM0335.

### 13. REFERENCES:

- 1. Bates T. A review of local radiotherapy in the treatment of bone metastases and cord compression. Int J Radiat Oncol Biol Phys 1992; 23:217-221
- 2. Maher EJ. The use of palliative radiotherapy in the management of breast cancer. Eur J Cancer 1992; 28:706-710.
- 3. Ratanatharathorn, Powers, Moss et al. Bone metastases: review and critical analysis of random allocation trials of local field treatment. Int. J. Radiat Oncol Biol Phys. 1994; 44:1-18.
- 4. McQuay, Collins, Carroll et al. Radiotherapy for the palliation of painful bone metastases. In: The Cochrane Library. 2002, Issue 1. Oxford: Update Software.
- 5. Wu, Wong, and Johnston et al. Meta-analysis of dose-fractionation radiotherapy trials for the palliation of painful bone metastases. Int. J. Radiat. Onc. Bio. Phys. 2003: Vol 55(3), pp.594-605, 2003.
- 6. Hartsell, Scott, Bruner, et al. Randomized trial of short versus long-course radiotherapy for palliation of painful bone metastases. JNCI. 2005; 97(11): 798-804.
- 7. Roos, Turner, O'Brien, et al. Randomized trial of 8 Gy in 1 versus 20 Gy in 5 fractions of radiotherapy for neuropathic pain due to bone metastases (TROG 96.05). Radiotherapy and Oncology. 2005; 75: 54-63.

- 8. Sze WM, Shelley MD, Wilt TJ, Mason MD. Palliation of Metastatic Bone Pain: Single fraction vs Multifraction Radiotherapy-A systematic Review of Randomized trials. Clinical Oncology. 2003; 15: 345-352.
- 9. Gaze MN, Kelly CG, Kerr GY, et al. Pain relief and quality of life following radiotherapy for bone metastases: a randomized trial of two fractionation schedules. Radiother Oncol. 1997; 45: 109-16.
- 10. Kagei K, Suzuki K, Shirato H, et al. A randomized trial of single and multifraction radiation therapy for bone metastasis: a preliminary report. Japan J Cancer Clin. 1990;36: 2553-8.
- 11. Ryu S, Jin R, Jin JJ, et al. Pain Control by Image-guided Radiosurgery for Solitary Spinal Metastases. J Pain Symp Manage. 2008; 35: 292-298.
- 12. Gerzten PC, Burton SA, Ozhasoglu C, et al. Radisurgery for the treatment of renal cell carcinoma. J Neurosurg Spine. 2005; 3(4): 288-295.
- 13. Garg AK, Shiu AS, Yang J. Phase I/II Trial of Single-session Stereotactic Body Radiotherapy for Previously Unirradiated Spinal Metastases. Cancer. 2012 Oct 15;118(20):5069-77
- 14. Korn EL, Freidlin B, Abrams JS, Halabi S. Design issues in randomized phase II/III trials. J Clin Oncol. 2012 Feb 20;30(6):667-71.
- 15. Bone Pain Trial Working Party. 8 Gy single fraction radiotherapy for the treatment of metastatic skeletal pain: randomized comparison with a multifraction schedule over 12 months of patient follow-up. Radiotherapy and Oncology. 1999;52:111-121.
- 16. Rubinstein LV, Korn EL, Freidlin B, Hunsberger S, Ivy SP, Smith MA. Design issues of randomized phase II trials and a proposal for phase II screening trials. J Clin Oncol 2005;23:7199-7206.
- 17. Thall PF, Simon RM, Estey EH. Bayesian sequential monitoring designs for single-arm clinical trials with multiple outcomes. Stat Med. 1995 Feb 28;14(4):357-79.
- 18. Gooley TA, Leisenring W, Crowley J, and Storer BE. Estimation of failure probabilities in the presence of competing risks: new representations of old estimators. Statistics in Medicine. 1999; 18:695-706.
- 19. Fine JP, Gray RJ. A proportional hazards model for the subdistribution of a competing risk. Journal of the American Statistical Association 1999;94:496-509.
- 20. Kaplan EL and Meier P. Nonparametric estimation from incomplete observations. Journal of the American Statistical Association 1958; 53:457-481.
- 21. Cox DR. Regression models and life tables (with discussion). Journal of the Royal Statistical Society B 1972; 34:187-220.
- 22. Paul A. Harris, Robert Taylor, Robert Thielke, Jonathon Payne, Nathaniel Gonzalez, Jose G. Conde. Research electronic data capture (REDCap) A metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform, 2009. 42(2):377-81.

# 14. TABLE A: PATIENT ASSESSMENT CHECKLIST

| Time | Н&Р | СВС | X-ray,<br>CT,<br>MRI,<br>bone<br>scan* | Path<br>Dx | MDASI<br>Survey | Phone<br>call<br>follow-<br>up | Toxicity/AE assessment |
|---|---|---|---|---|---|---|---|
| Pre-RT | Х | Х | Х | Х | Х | | Х |
| Within 7-10 days post | | | | | X | Х | |
| 1 month post XRT <sup>2</sup> | | | | | Х | Х | |
| 3 month f/u <sup>1</sup> | | | х | | Х | | Х |
| 6 month<br>f/u <sup>1</sup> | | | х | | X | | Х |
| 9 month<br>f/u <sup>1</sup> | | | Х | | х | | Х |
| 12 month<br>f/u <sup>1</sup> | | | X | | Х | | Х |
| 3-6 month interval thereafter (until death) | | | X | | X | | X |

<sup>\*</sup>Per standard of care

<sup>&</sup>lt;sup>2</sup> Within +/- 1 week

| Time | H&P | СВС | X-ray,<br>CT,<br>MRI,<br>bone<br>scan* | Path<br>Dx | MDASI<br>Survey | Narcotic/<br>Opioid/<br>NSAID<br>use | Toxicity/AE<br>assessment |
|---|---|---|---|---|---|---|---|
| Pre-RT | X | Χ | Χ | X | X | X | X |
| Within 7-14 days post start of XRT by phone | | | | | X | X | x |
| 1 month post start of<br>XRT by phone <sup>2</sup> | | | | | Х | Х | Х |
| 3 month f/u <sup>1</sup> | | | X | | Х | X | X |

<sup>&</sup>lt;sup>1</sup> Within +/- 4 weeks

| 6 month f/u <sup>1</sup> | Х | Х | Х | Х |
|---------------------------------------------|---|---|---|---|
| 9 month<br>f/u <sup>1</sup> | X | X | X | X |
| 12 month f/u <sup>1</sup> | Х | X | X | X |
| 3-6 month interval thereafter (until death) | Х | х | Х | х |

<sup>\*</sup>Per standard of care

15. APPENDIX A: NCI CTCAE version 4.03

16. APPENDIX B: The M.D. Anderson Symptom Inventory (MDASI) survey

<sup>&</sup>lt;sup>1</sup> Within +/- 4 weeks

<sup>&</sup>lt;sup>2</sup> Within +/- 1 week